CLINICAL TRIAL: NCT02788227
Title: A Multicenter Study of the Immunogenicity of Recombinant Vesicular Stomatitis Vaccine for Ebola-Zaire (rVSVdeltaG-ZEBOV GP) for Pre-Exposure Prophylaxis in Individuals at Potential Occupational Risk for Ebola Virus Exposure (PREPARE)
Brief Title: Immunogenicity of Recombinant Vesicular Stomatitis Vaccine for Ebola-Zaire (rVSV[Delta]G-ZEBOV-GP) for Pre-Exposure Prophylaxis (PREP) in People at Potential Occupational Risk for Ebola Virus Exposure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 160053; 16-I-0053
Record Dates: First submitted 2016-05-28; First posted 2016-06-02 (Estimated); Last update posted 2025-07-01 (Actual); Status verified 2025-06-18

CONDITIONS: Healthy Volunteers
Keywords: Ebola Vaccine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Boosted Group (Experimental): Group randomized at Month 18 to receive booster vaccination
  Interventions: Biological: rVSV-Zebov GP vaccine
- Non-boosted Group (Experimental): Group randomized to 'no booster' at Month 18
  Interventions: Biological: rVSV-Zebov GP vaccine

INTERVENTIONS:
Biological: rVSV-Zebov GP vaccine — primary vaccination for all participants, one-to-one randomization at Month 18 to receive booster vaccination or no booster.

SUMMARY:
Background:

The Ebola virus causes a severe disease. It can be fatal. The usual incubation period after being exposed is 2 to 21 days. There is no approved treatment for Ebola infection. There is also no vaccine to prevent infection either before or after exposure. Researchers want to test an Ebola vaccine. They want to give it to people before they are exposed to the virus in order to prevent the disease.

Objectives:

To see how long-lasting and effective the vaccine rVSV[delta]G -ZEBOV-GP (V920) is at preventing Ebola.

Eligibility:

Healthy adults at risk of exposure to the Ebola virus at work through lab or clinical contact.

Design:

Participants will be screened with medical history, physical exam, and blood tests.

Participants will get the study vaccine. It will be injected into their upper arm.

Participants will be monitored closely for at least 30 minutes. They will get a diary card to record any symptoms they have from the vaccine for up to 14 days.

Participants will have study visits at 1, 3, and 6 months after they get the vaccine, then every 6 months (that is, at months 12, 18, 19, 24, 30, and 36 of study) for a total of 36 months.

Eighteen months after they join the study, participants will be randomly assigned to one of two groups. One group will get a second (or booster ) dose of the vaccine. The other group will not get a second dose.

This study lasts 36 months. In December 2024, the study was approved to re-enroll up to 30 participants from the primary cohort to check longer-term immune response to the study vaccine beyond 36 months.

DETAILED DESCRIPTION:
Between 1994 and the present, there have been multiple Ebolavirus outbreaks affecting mostly central Africa. However, the 2014/2015 West African outbreak significantly exceeds all previous outbreaks in geographic range, number of individuals affected, and in disruption of typical activities of civil society.

This protocol is a multi-center study to evaluate the durability of the immune response following the open label administration of the rVSVdeltaG-ZEBOV-GP vaccine (V920) as pre-exposure prophylaxis for adults who have an occupational risk for potential exposure to Ebola virus. The vaccine uses a live replicating vesicular stomatitis virus (VSV) replacing the gene encoding the G envelope glycoprotein with the gene encoding the envelope glycoprotein from the Zaire strain of Ebola (rVSVdeltaG-ZEBOV-GP also known as V920).

All subjects will receive a single dose of rVSVdeltaG-ZEBOV-GP (>=7.2 x 10^7 pfu) on Day 0. We will collect adverse events after vaccination and at Month 1 and Month 19, serious adverse events (SAE) for the duration of the study, and assess the immune response at Months 1, 3, 6, 12, 18, 19, 24, 30, and 36.

A single booster immunization with the same dose of study vaccine as the primary dose (>=7.2 x 10^7 pfu/mL) will be given to those randomized at month 18 to the booster arm of the trial. However, if at any time during the observation period antibody levels fall below a predefined seroprotective threshold (yet to be defined in parallel or newly planned studies), a booster will be offered to those who have not previously received a booster injection.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Adults age >=18 years.
2. Signed informed consent for the trial.
3. At risk of occupational exposure to Ebola virus through laboratory, clinical contact, or field work, in the judgment of the investigator.
4. Females of childbearing potential must be willing to use effective methods of contraception, from at least 30 days prior to vaccination through 1 month following vaccination/booster, which would include:

   * oral contraceptives, either combined or progestogen alone
   * injectable progestogen
   * implants of etenogestrel or levonorgestrel
   * oestrogenic vaginal ring
   * percutaneous contraceptive patches
   * intrauterine device or intrauterine system
   * committed to abstinence from potentially reproductive sexual contact [i.e. will NOT engage in heterosexual intercourse where both partners are capable of reproduction]
   * surgical sterilization
   * male condom combined with a spermicide
5. All males must be willing to use effective methods of contraception for at least 1 month following vaccination/booster, which would include:

   * surgical sterilization
   * male condom combined with a spermicide
6. Willing to minimize blood and body fluid exposure to others for at least 14 days after vaccination/booster. This includes:

   * Use of effective barrier prophylaxis, such as latex condoms, during any sexual interaction (regardless of childbearing status or sexual orientation)
   * Avoiding the sharing of needles, razors, eating utensils, drinking from the same cup, or toothbrushes
   * Avoiding open-mouth kissing
   * Use of universal precautions in the health-care setting
7. Agrees not to receive another investigational agent between vaccination and the Month 1 study visit (and booster and Month 19 study visit).
8. Willing to forgo blood donation for one year from vaccination/booster.
9. Willing to accept randomization (boost versus no boost) at month 18 visit.

EXCLUSION CRITERIA:

1. Any condition that would limit the ability of the participant to meet protocol requirements or would place the participant at unreasonable risk. Examples include:

   * Clinically significant medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health, per the investigator. A clinically significant condition or process includes but is not limited to:

     1. A process that would adversely affect the systemic immune response
     2. A process that would require medication that might adversely affect the systemic immune response
     3. Any contraindication to repeated injections or blood draws
     4. A condition that requires active medical intervention or monitoring to avert grave danger to the participant's health or well-being during the study period
     5. A condition or process for which signs or symptoms could be confused with reactions to vaccine
   * Presence of any pre-existing illness or clinical history that, in the opinion of the investigator, would place the participant at an unreasonably increased risk through participation in this study. This includes but is not limited to:

     1. Active malignancy
     2. History of Guillain-Barre Syndrome
     3. History of neurological disorder that may increase risk (history of encephalitis, stroke, or seizure)
     4. Active autoimmune disorder requiring systemic immunosuppressive treatment
   * Any concomitant medication for which reported side effects or adverse events, in the judgment of the investigator, may interfere with assessment of safety.
   * Subjects who, in the judgment of the investigator, will be unlikely or unable to comply with the requirements of this protocol.
2. Pregnant or breast feeding (must have negative serum or urine pregnancy test on the day of vaccination, prior to vaccination)
3. Known allergy to the components of the rVSVdeltaG-ZEBOV-GP vaccine (V920) vaccine product (VSV, albumin, tris).
4. History of severe local or systemic reactions to any vaccination.
5. Received an investigational drug within 5 half-lives or 30 days, whichever is longer, prior to vaccination (Day 0)/booster (Month 18).
6. Received killed vaccines 14 days before, or intention to receive within 7 days following, vaccination (Day 0)/booster (Month 18).
7. Received live virus vaccines within 30 days before, or intention to receive live virus vaccines within 30 days following, vaccination (Day 0)/booster (Month 18).
8. Received immunoglobulins and/or any blood products within the 120 days preceding vaccination (Day 0)/booster (Month 18).
9. Received allergy treatment with antigen injections within 30 days before vaccination (Day 0)/booster (Month 18).
10. Clinical evidence (e.g. oral temp >38 degrees Celsius, systemic symptoms) of a systemic infection or other acute intercurrent illness at the proposed time of vaccination (Day 0)/booster (Month 18).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2016-10-14 (Actual); Primary Completion 2025-06-17 (Actual); Study Completion 2025-06-17 (Actual)

PRIMARY OUTCOMES:
Comparison of antibody titer levels between the boosted vs non-boosted groups | Month 36
  Titer levels in EU/mL

CONTACTS AND LOCATIONS:
Overall Officials: Susan L Moir, Ph.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
Individual (coded with Participant ID only) data and antibody titer levels are shared with the University of Minnesota Data Center for statistical evaluation. The study team is blinded to the titers after Month 18 timepoint for all subjects. When the endpoint of the study is reached (i.e. when a statistically significant number of subject have reached Month 36/end-of-study), data will likely be shared with other study sites.

REFERENCES:
- [Background] Regules JA, Beigel JH, Paolino KM, Voell J, Castellano AR, Hu Z, Munoz P, Moon JE, Ruck RC, Bennett JW, Twomey PS, Gutierrez RL, Remich SA, Hack HR, Wisniewski ML, Josleyn MD, Kwilas SA, Van Deusen N, Mbaya OT, Zhou Y, Stanley DA, Jing W, Smith KS, Shi M, Ledgerwood JE, Graham BS, Sullivan NJ, Jagodzinski LL, Peel SA, Alimonti JB, Hooper JW, Silvera PM, Martin BK, Monath TP, Ramsey WJ, Link CJ, Lane HC, Michael NL, Davey RT Jr, Thomas SJ; rVSVDeltaG-ZEBOV-GP Study Group. A Recombinant Vesicular Stomatitis Virus Ebola Vaccine. N Engl J Med. 2017 Jan 26;376(4):330-341. doi: 10.1056/NEJMoa1414216. Epub 2015 Apr 1. PMID 25830322
- [Background] Agnandji ST, Huttner A, Zinser ME, Njuguna P, Dahlke C, Fernandes JF, Yerly S, Dayer JA, Kraehling V, Kasonta R, Adegnika AA, Altfeld M, Auderset F, Bache EB, Biedenkopf N, Borregaard S, Brosnahan JS, Burrow R, Combescure C, Desmeules J, Eickmann M, Fehling SK, Finckh A, Goncalves AR, Grobusch MP, Hooper J, Jambrecina A, Kabwende AL, Kaya G, Kimani D, Lell B, Lemaitre B, Lohse AW, Massinga-Loembe M, Matthey A, Mordmuller B, Nolting A, Ogwang C, Ramharter M, Schmidt-Chanasit J, Schmiedel S, Silvera P, Stahl FR, Staines HM, Strecker T, Stubbe HC, Tsofa B, Zaki S, Fast P, Moorthy V, Kaiser L, Krishna S, Becker S, Kieny MP, Bejon P, Kremsner PG, Addo MM, Siegrist CA. Phase 1 Trials of rVSV Ebola Vaccine in Africa and Europe. N Engl J Med. 2016 Apr 28;374(17):1647-60. doi: 10.1056/NEJMoa1502924. Epub 2015 Apr 1. PMID 25830326
- [Derived] Davey RT Jr, Collins GL, Rouphael N, Poliquin G, McConnell R, Grubbs G, Moir SL, Langley JM, Teitelbaum M, Hewlett AL, McLellan SLF, Bhadelia N, Raabe VN, Mulligan MJ, Maljkovic Berry I, Dighero-Kemp B, Kurtz JR, Hensley LE, Dozier NCE, Marron LCB, DuChene A, Kuhn JH, Brown SK, Khurana S, Lane HC, Neaton JD. Safety and immunogenicity of a delayed booster dose of the rVSVDeltaG-ZEBOV-GP vaccine for prevention of Ebola virus disease: a multicentre, open-label, phase 2 randomised controlled trial. Lancet Microbe. 2024 Nov;5(11):100923. doi: 10.1016/S2666-5247(24)00163-0. Epub 2024 Oct 4. PMID 39374605
- [Derived] Raabe V, Lai L, Morales J, Xu Y, Rouphael N, Davey RT, Mulligan MJ. Cellular and humoral immunity to Ebola Zaire glycoprotein and viral vector proteins following immunization with recombinant vesicular stomatitis virus-based Ebola vaccine (rVSVDeltaG-ZEBOV-GP). Vaccine. 2023 Feb 17;41(8):1513-1523. doi: 10.1016/j.vaccine.2023.01.059. Epub 2023 Jan 31. PMID 36725433
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2016-I-0053.html